## "AUDITORY BRAIN TRAINING TO ENHANCE SATISFACTION AND USAGE OF NEW HEARING AIDS BY OLDER ADULTS"

## NCT04230876

Document Date/Version: 6/15/22

Data will be analyzed with Repeated measures ANOVA to assess the effect of training on use time, changes in speech perception, and subjective changes indicated by the questionnaire rating-scale responses. Repeated measures will compare changes in outcome measures for the time spent during training to changes during the time spent not in the training. The numbers of participants in each group was determined based on effect sizes for the COSI in Tye-Murray et al. (2016), who found differences post-training using the same primary outcome measure, a similar training schedule and similar methods proposed here. We determined the power to detect an effect size for differences as large as or larger than in Tye-Murray et al. (mean = .733, SD = .783) with an alpha level of .05 will approach .95 using a one-tailed test for the within-subjects comparisons.